CLINICAL TRIAL: NCT06137885
Title: Registry-based Cardiovascular Quality Improvement Research (RESCUER)
Brief Title: REgiStry-based Cardiovascular qUality improvEment Research
Acronym: RESCUER
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: RESCUER-2022
Record Dates: First submitted 2023-10-20; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Percutaneous Coronary Intervention; Heart Failure; Cardiometabolic Syndrome; Structural Heart Abnormality
Keywords: Cardiovascular Diseases; Registry; Cardiac rehabilitation; Active device surveillance; Multi-omics
MeSH Terms: conditions — Heart Failure; Metabolic Syndrome; Cardiovascular Diseases | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, urine, saliva, feces, cardiac tissue ()
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PCI group: Patients who received percutaneous coronary intervention (PCI) at the Department of cardiology of Peking University Third Hospital will be included in the PCI group.
  Interventions: Behavioral: Cardiac rehabilitation; Other: Active post-market surveillance of devices; Other: Multi-omics approach to precision medicine; Other: The prescription pattern analysis
- Heart failure group: Patients with heart failure who hospitalized at the Department of cardiology of Peking University Third Hospital will be included in the heart failure group.
  Interventions: Behavioral: Cardiac rehabilitation; Other: Active post-market surveillance of devices; Other: Multi-omics approach to precision medicine; Other: The prescription pattern analysis
- Cardiometabolic syndrome group: Patients with cardiometabolic syndrome who hospitalized at the Department of cardiology of Peking University Third Hospital will be included in the cardiometabolic syndrome group.
  Interventions: Behavioral: Cardiac rehabilitation; Other: Multi-omics approach to precision medicine; Other: The prescription pattern analysis
- Structural heart disease group: Patients with structural heart disease who hospitalized at the Department of cardiology of Peking University Third Hospital will be included in the structural heart disease group.
  Interventions: Behavioral: Cardiac rehabilitation; Other: Active post-market surveillance of devices; Other: Multi-omics approach to precision medicine; Other: The prescription pattern analysis

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Cardiac rehabilitation is a comprehensive model of care involving prescribed exercise, medication management, lifestyle modification, and psychosocial counseling to help people with heart diseases resume and enhance their psychosocial and vocational status.
Other: Active post-market surveillance of devices — Active post-market surveillance of devices is an essential and ongoing process that involves systematic monitoring and assessment of medical devices once they are available on the market. It involves continuous data collection and analysis, early detection of issues, risk assessment, compliance with regulatory requirements, adaptive decision-making, and transparent communication with healthcare professionals and patients.
  Groups: Heart failure group; PCI group; Structural heart disease group
Other: Multi-omics approach to precision medicine — Multi-omics analysis refers to the collective analysis of extensive biological data from multiple omics sources to gain a holistic understanding of an individual's health status, disease susceptibility, and response to therapies. By considering a broad spectrum of genetic and molecular information, multi-omics precision medicine aims to deliver more accurate diagnoses, predict disease risks, select optimal treatment options, and monitor therapeutic responses with a high degree of specificity, ultimately improving patient outcomes and minimizing adverse effects.
Other: The prescription pattern analysis — The prescription pattern analysis refers to the systematic examination and evaluation of the types, dosages, frequencies, and trends in medications prescribed to patients with cardiovascular conditions. By scrutinizing prescription patterns, researchers and healthcare professionals can identify prevalent medications, assess adherence to treatment guidelines, uncover potential gaps or areas for improvement in patient care, and gain insights into the evolving landscape of cardiovascular therapies.

SUMMARY:
The goal of this registry-based observational study is to establish a comprehensive management plan, which focus on medical therapy, cardiac rehabilitation and active post-market surveillance of medical devices, in patients with cardiovascular diseases (CVD). Patients with CVD mainly refers to four groups of patients：1) post-percutaneous coronary intervention (post-PCI) patients; 2) patients with heart failure (HF); 3) patients with cardiometabolic diseases (CMD); 4) patients with structural heart disease (SHD), and the detailed definition of each group can be found in "Eligibility" section. The main questions this study aims to answer are:

* the effectiveness of exercise-based cardiac rehabilitation in improving cardiac function, reducing CVD recurrence and mortality, and promoting quality of life for patients with CVD;
* the feasibility of registry-based active post-market surveillance of high-risk medical devices used in cardiovascular surgeries, such as PCI, heart valve replacement, and cardiac resynchronization therapy (CRT);
* the utilization of multiomics datasets to identify and dissect cardiovascular heterogeneity in both healthy and diseased populations and to guide precision medicine in patients with CVD;
* the analysis and evaluation of the prescription patterns and drug response in patients with CVD.

DETAILED DESCRIPTION:
This is a long-term registry, which will continuously enroll patients and approximately 2000 subjects will be enrolled during the first phase.

Primary analyses may include, but will not be limited to, the following: incidence of MACE, procedural complications, and changes in patients' quality of life. Descriptive statistics will be used for baseline, procedure and follow-up data collected through the study.

Each patient will be followed for a period of two years after enrollment according to the schedule and standard practice at Peking University Third Hospital. The follow-up schedule is 2 weeks, 1 month ( additional for HF group), 3 months, 6 months, 12 months, 24 months after discharge. For patients who miss a follow-up visit, a contact (e.g. phone call) will ensure capture of the endpoint related information. In addition, all fatal events will be tracked from the death registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with cardiovascular diseases who are hospitalized at the Department of Cardiology of Peking University Third Hospital after April 24th, 2023;
* Patients meet the following disease definitions:

  1. PCI group: Patients underwent percutaneous coronary intervention (PCI) or coronary angiography;
  2. HF group: Patients diagnosed with heart failure;
  3. Cardiometabolic Disease (CMD) group: Patients with cardiovascular disease (primarily including coronary artery disease, peripheral artery disease, and aortic disease) and coexisting metabolic disorder (defined as obesity [BMI≥28 kg/m^2], prediabetes and diabetes, hypertension, hyperlipidemia, thyroid dysfunction, and non-alcoholic fatty liver disease);
  4. Structural Heart Disease (SHD): Patients with structural heart disease, including

     * Congenital heart diseases (such as ventricular septal defect, atrial septal defect, patent ductus arteriosus, tetralogy of Fallot, etc.);

       * Heart valve diseases (mitral valve, tricuspid valve, aortic valve, pulmonary valve, etc.);

         * Cardiomyopathies (hypertrophic cardiomyopathy, dilated cardiomyopathy, etc.);

           * Conditions associated with other diseases or acquired structural abnormalities of the heart (ventricular septal perforation, ventricular aneurysm, iatrogenic atrial septal defect, etc.);

             * Conditions resulting from other diseases that cause abnormal heart function, which can be corrected by altering cardiovascular structure (such as left atrial appendage dysfunction caused by atrial fibrillation, abnormal cardiac function caused by heart failure);

               * Others: Intracardiac thrombosis, cardiac tumors, pericardial diseases, etc.

Exclusion Criteria:

* patients with no informed consent form (ICF) or who withdraw ICF；
* patients with cognitive impairment or those unable to complete the questionnaire required in the study;
* patient who is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 4 groups of adult patients with cardiovascular diseases (PCI group, HF group, CMD group, SHD group) who are hospitalized at the Department of Cardiology of Peking University Third Hospital after they provide the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
MACE (PCI group and CMD group) | Assessed at each scheduled follow-up and all fatal events will be tracked from the death registry
  Major Adverse Cardiovascular Events (MACE): non-fatal myocardial infarction, non-fatal stroke, unstable angina, and all-cause mortality.
Composite Endpoint：cardiovascular death+ HF-related rehospitalization. | Assessed at each schedule follow-up and all fatal events will be tracked from the death registry
  Primary outcome for HF group
Composite Endpoint：cardiovascular death+ rehospitalization. | Assessed at each scheduled follow-up and all fatal events will be tracked from the death registry
  Primary outcome for SHD group

SECONDARY OUTCOMES:
3-point MACE (PCI group and CMD group) | Assessed at each scheduled follow-up and all fatal events will be tracked from the death registry
  3 point MACE: non-fatal myocardial infarction, non-fatal stroke, and cardiovascular death.
Cardiovascular death (HF group) | Assessed at each scheduled follow-up and all fatal events will be tracked from the death registry
  Cardiovascular death refers to a type of death that occurs as a result of diseases or conditions affecting the cardiovascular system, which includes the heart and blood vessels.
HF-related rehospitalization (HF group) | Assessed at each scheduled follow-up
  HF-related rehospitalization refers to the situation where an individual who has previously been hospitalized for heart failure (HF) experiences a recurrence or worsening of their heart failure symptoms and needs to be readmitted to the hospital for further medical treatment and care.
Composite outcome of bleeding and transfusion | Assessed at each scheduled follow-up and during hospitalization
  Bleeding and transfusion are defined using the Bleeding Academic Research Consortium (BARC) categories.
Composite outcome of in-hospital device-related adverse events | In hospital
  In-hospital device-related adverse event outcomes are defined as device embolization, device fracture, device thrombosis, device displacement, heart arrest, and cardiac perforation.
Composite outcome of long-term device-related adverse events | Assessed at each scheduled follow-up
  Long-term device-related adverse event outcomes are defined as device embolization and device thrombosis.
Changes in patients' peak oxygen uptake | Assessed at each each scheduled follow-up
  The peak oxygen uptake is measured by the cardiopulmonary exercise test (CPET).
Changes in health related quality of life scores reported by participants via EuroQol-5 dimensions (EQ-5D) questionnaire | Assessed at each scheduled follow-up
  Changes in patients' quality of life scores are measured by EQ-5D questionnaire.
Changes in health related quality of life scores reported by participants via Kansas City Cardiomyopathy Questionnaire (KCCQ) (for HF group and SHD group) | Assessed at each scheduled follow-up
  The KCCQ measures symptoms, physical and social limitations, and quality of life in patients with heart failure and structural heart diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Yida Tang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data, analytic methods, and study materials will not be made available immediately to other researchers. Request to get these materials can be sent to the study PI, and we will provide them to vetted and qualified applicants.